CLINICAL TRIAL: NCT03503097
Title: GENTleMEN: Genetic Testing for Men With Metastatic Prostate Cancer
Brief Title: Genetic Testing for Men With Metastatic Prostate Cancer
Acronym: GENTleMEN
Status: Terminated | Type: Observational
Why Stopped: Study closed to accrual before meeting enrollment goal due to end of funding.
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 9831; NCI-2018-00533 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9831 (Other: Fred Hutch/University of Washington Cancer Consortium); RG1001545 (Other: Fred Hutch/University of Washington Cancer Consortium); 5P50CA097186-17 (NIH)
Record Dates: First submitted 2018-04-11; First posted 2018-04-19 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Prostate Carcinoma; Stage IV Prostate Cancer AJCC v8; Stage IVB Prostate Cancer AJCC v8
Keywords: Prostate cancer; metastatic; genetic testing; cancer risk; BRCA1; BRCA2
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — Genetic Counseling; Genetic Testing; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ancillary-Correlative (questionnaires, Color kit, counseling): Participants receive web-based or hard-copy questionnaires and saliva collection kits via mail or in person. Participants also provide saliva samples to be mailed back to Color Genomics for genetic testing once complete. Participants then receive phone-based genetic counseling if they are identified to have an inherited mutation in a DNA repair gene. All participants have access to phone-based genetic counseling whether or not they are not found to have a mutation.
  Interventions: Procedure: Biospecimen Collection; Other: Genetic Counseling; Other: Genetic Testing; Other: Laboratory Biomarker Analysis; Behavioral: Questionnaire

INTERVENTIONS:
Procedure: Biospecimen Collection — Provide saliva samples
Other: Genetic Counseling — Undergo counseling
Other: Genetic Testing — Undergo genetic testing
  Other Names: genetic analysis; Genetic Examination; Genetic Test
Other: Laboratory Biomarker Analysis — Correlative studies
Behavioral: Questionnaire — Complete questionnaire
  Other Names: Questionnaires

SUMMARY:
This research study provides genetic testing to men with prostate cancer that has spread to other parts of the body (metastatic prostate cancer) and will look for inherited genetic mutations in about 30 cancer-risk genes. The researchers seek to learn about the participant's opinions and concerns about genetic testing, to determine if this is an acceptable way to deliver testing and to potentially help guide the participant's treatment. Neither treatment nor any decisions related to treatment will take place on this study, but researchers will share each participant's genetic testing results with that participant.

DETAILED DESCRIPTION:
OUTLINE:

Participants receive web-based or hard-copy questionnaires and saliva collection kits via mail or in person. Participants also provide saliva samples to be mailed back to Color Genomics for genetic testing once complete. Participants then receive phone-based genetic counseling if they are identified to have an inherited mutation in a deoxyribonucleic acid (DNA) repair gene. All participants have access to phone-based genetic counseling whether or not they are not found to have a mutation.

After study completion, participants are followed up at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form (ICF) providing agreement for germline genetic testing, use and release of health and research trial information
* Documented evidence of metastatic prostate cancer;

  * Oncologist note within 4 months
  * All computed tomography (CT), bone, positron emission tomography (PET) scan reports within 12 months
  * All prostate-specific antigen (PSA) values within 12 months
  * All available pathology reports from diagnosis, prostatectomy, and/or metastatic biopsy
* Willingness to provide basic demographic information, family cancer history, and treatment history
* Willingness and ability to complete patient reported outcomes questionnaire (on-line or hard copy) at enrollment, and at 6-month follow-up
* Willingness and ability to provide saliva sample

Exclusion Criteria:

* Unable or unwilling to provide all of the necessary information for eligibility, e.g. decisionally impaired
* Incomplete inclusion criteria
* Study team members

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with metastatic prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 799 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2024-08-21 (Actual); Study Completion 2025-09-17 (Actual)

PRIMARY OUTCOMES:
Frequency of pathogenic germline homologous recombination (HR) variants in men with metastatic prostate cancer (mPC) | From the start of study up to 3 years
  Frequency to be determined by genetic testing on saliva samples for inherited mutations in cancer risk genes such as BRCA2, BRCA1, ATM, and others in metastatic prostate cancer.
Patient reported outcome measures associated with genetic testing in men with mPC | From the time of enrollment up to 6-month follow-up
  Outcome measures to be defined by patient reported outcomes questionnaire (on-line or hard copy) at enrollment, and at 6-month follow-up.
Utility of family history to enrich screening of participants with mPC for germline homologous recombination deficiency (HRD) variants defined by collection of information about research participants' family history | From the start of study up to 3 years
  To be determined by collection of information about research participants' family history that includes cancer history (diagnosis, age of onset, treatment, etc.) but will not include identifiers of family members. This information will be used to examine which self-reported family history criteria may be associated with identification of cancer predisposition syndrome.
Identification of a cohort of men with prostate cancer and inherited HRD mutations | From the start of study up to 3 years
  Identification to be determined through the Washington state cancer registry, through mail-out to all urologists and medical oncologists in the state of Washington, and through the Seattle Cancer Care Alliance Network sites. In addition, web-based advertising and recruiting will occur more broadly through the U.S., including at partnering sites.

CONTACTS AND LOCATIONS:
Overall Officials: Heather H. Cheng, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States